CLINICAL TRIAL: NCT01864811
Title: The Efficacy of Constraint Induced Movement Therapy for Babies (Baby-CIMT) in Infants Below 12 Month With Risk of Developing Unilateral Cerebral Palsy, a Study Protocol of a Randomized Controlled Trial
Brief Title: Effect of Baby-CIMT in Infants Younger Than 12 Months
Acronym: B-CIMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ann-Christin Eliasson, professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFO-V4072/2012; 2011-1522-81929-42 (Other Grant/Funding Number: Swedish Research Counsil)
Record Dates: First submitted 2013-05-22; First posted 2013-05-30 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Cerebral Palsy; Hemiplegia; Children
Keywords: infants; unilateral cerebral pares; hand function; early intervention; constraint induced movement therapy
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baby-CIMT (Experimental): The infants will be prevented from using the preferred hand while the other hand will be trained using amusing and easily handled toys.
  Interventions: Behavioral: Baby-CIMT
- baby-massage (Experimental): The infants will receive baby massage
  Interventions: Behavioral: Baby-Massage

INTERVENTIONS:
Behavioral: Baby-CIMT — Baby-CIMT is a very much modified model of constraint induced movement therapy for infants. It is developed to suit small children and their needs of stimulation. The infant should wear a comfortable glove on the less affected hand, while stimulating the use of the affected hand 30 minutes per day during 2 periods of 6-weeks training before 12 month. The hand training provides the baby with amusing and easily handled toys.
  Other Names: Constraint Induced Movement therapy
  Arms: Baby-CIMT
Behavioral: Baby-Massage — For baby massage, there will be a special instructional course by a health professional certified for baby massage. Massage should be given every day during 2 periods of 6 weeks. Families will be responsible for the massage.
  Arms: baby-massage

SUMMARY:
A randomized control trial investigating if an early intervention program of modified Constraint Induced Movement Therapy for babies, Baby-CIMT, performed before 12 months of age will improve hand function in children with risk for developing cerebral palsy.

DETAILED DESCRIPTION:
The investigators hypothesis is that Baby-CIMT including intensive specific task oriented training is more preferable than general stimulation which is the assumption for baby massage used in the control group. The intervention protocol is developed at Astrid Lindgren Children hospital, Stockholm Sweden.

ELIGIBILITY:
Inclusion Criteria:1. A neonatal history of different origin of events affecting the brain, preterm children with predominantly unilateral hemorrhage, venous infarction or with matter lesion or pre, perinatal or early postnatal stroke or Infants referred to the hospital/rehabilitation centers/specialists with signs of asymmetries before 8 month of age, likely to be diagnosed with unilateral cerebral palsy at later age.

Recruitment criteria of child characteristics

* Age can vary, earliest at 3 months of age and at the latest at 8 months
* Sign of asymmetries from mild to clear and severe asymmetries,

Exclusion Criteria:

Severe visual impairment Seizures not controlled by drugs Not unilateral CP at 12 month

Ages: 3 Months to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Hand Assessment for Infants (HAI) | 12 month post term age
  Hand Assessment for Infants (HAI) identify and measure upper limb asymmetry and general manual development from 3-12 month in children at risk of developing cerebral palsy.Even though our Primary Outcome Measure is when children are at one year post term age, we are going to publish results from assessments at earlier ages to measure changes after each intervention period.

SECONDARY OUTCOMES:
Alberta Motor Infant Scale | Baseline and12 months post term age
  Identification of infants who are delayed or deviant in motor development and evaluation of motor development over time. Identifies gross motor performance of an infant compared to norm- referenced sample.

OTHER OUTCOMES:
To Be a Parent: a questionary | 12 monts post preterm
  16 statement as both parents has to fill in. they have to agree on the statement based on a 6-grading scale

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Christin Eliasson, professor, Principal Investigator — Department of Women's and Children's Health, Karolinska Univeristy
Locations (1):
- Astrid Lindgren Children Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Greaves S, Imms C, Krumlinde-Sundholm L, Dodd K, Eliasson AC. Bimanual behaviours in children aged 8-18 months: a literature review to select toys that elicit the use of two hands. Res Dev Disabil. 2012 Jan-Feb;33(1):240-50. doi: 10.1016/j.ridd.2011.09.012. Epub 2011 Oct 11. PMID 22093670